CLINICAL TRIAL: NCT05241145
Title: A Randomized, Controlled, Double-Masked Evaluation of the Safety and Preliminary Efficacy of IVMED-80 on Keratoconus Progression
Brief Title: Safety and Preliminary Efficacy of IVMED-80 Eye Drops in Keratoconus Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: iVeena Delivery Systems, Inc. (Industry)
Collaborators: Codet Vision Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IVNA 17-02
Record Dates: First submitted 2022-02-05; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Keratoconus; Corneal Ectasia
Keywords: Keratoconus; Corneal Ectasia; Copper; Micronutrients; Eye drops; Topical Therapy
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Intervention Model Description: This study used a three-arm, parallel design. Eligible study patients were randomly assigned to 1 of 3 treatment group following a 1:1:1 schedule.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigational products, IVMED-80 or Placebo (IVMED-80 vehicle solution) eye drops, were masked to all sponsor and site personnel with the exception of those directly involved with the production, labeling and shipping of product to the study sites. During the study, the identity of the test articles and randomization were not revealed. An unmasked study coordinator managed test article receipt, dispensing and inventory at the study site. Investigators who interacted with study patients to assess safety and efficacy were masked as to the identity of the test articles and treatment group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- IVMED-6Wk (Experimental): In Group 1 (IVMED-6Wk), patients instilled IVMED-80 eye drops into their study eye twice a day for 6 weeks and were followed for an additional 20 weeks without treatment (total 26 weeks)
  Interventions: Drug: IVMED-80
- IVMED-16Wk (Experimental): In Group 2 (IVMED-16Wk), patients instilled IVMED-80 eye drops into their study eye twice a day for 16 weeks and were followed for an additional 10 weeks without treatment (total 26 weeks)
  Interventions: Drug: IVMED-80
- Placebo (Placebo Comparator): In Group 3 (Placebo), patients instilled IVMED-80 vehicle solution eye drops into their study eye twice a day for 16 weeks and were followed for an additional 10 weeks without treatment (total 26 weeks)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: IVMED-80 — Good Manufacturing Practices-grade copper (ІІ) sulfate pentahydrate (CuSO4 #5H2O MW 249.69) was dissolved in a vehicle solution comprised of a balanced salt solution (BSS) with osmolality of approximately 500 mOsm/L. Copper sulfate was concentrated to 0.15 mg/mL. The drops were manufactured on prior to the study at a compounding pharmacy in Salt Lake City, Utah.
  Arms: IVMED-16Wk; IVMED-6Wk
Other: Placebo — This was identical to the IVMED-80 product, but without the active ingredient, copper sulfate.
  Other Names: IVMED-80 Vehicle
  Arms: Placebo

SUMMARY:
We investigated the use of a copper sulfate eye drop (IVMED-80) for the treatment of keratoconus. Preliminary laboratory data shows that the addition of copper sulfate increase crosslinking of the structural proteins of the cornea thereby halting the progressing corneal thinning and bulging seen in keratoconus. We conducted a Phase 1/2a study to evaluate the safety and preliminary efficacy of a 6-week and a 16-week regimen using IVMED-80 and studied its impact on ocular safety and the change/progression in patients' vision and clinical measurements.

DETAILED DESCRIPTION:
Standard Operating Procedures:

This study was designed to evaluate the safety and preliminary efficacy of IVMED-80 (0.15 mg/mL copper sulfate pentahydrate) in controlling the progression of corneal changes which typically occur in keratoconus patients.

This was a randomized, double-masked, placebo-controlled, and single-site clinical trial with eligible patients randomly assigned to one of three treatment groups:

* Group 1 (IVMED-6Wk) received topical copper sulfate eye drops 2x/day (BID) for 6 weeks and followed by an additional 20 weeks without treatment (total 26 weeks).
* Group 2 (IVMED-16Wk) received topical copper sulfate eye drops BID for 16 weeks and followed for an additional 10 weeks without treatment (total 26 weeks).
* Group 3 (Placebo) received IVMED-80 vehicle eye drops BID for 16 weeks and followed for an additional 10 weeks without treatment (total 26 weeks).

All patients were seen at Screening Visit, at Day 0 (Dispensing), and on Weeks 1, 3, 6, 12, 16, 21 and 26. In-office ophthalmology examinations used marketed medical diagnostic devices and routine clinical procedures. If a patient presents with two eyes meeting the eligibility criteria, the eye with the worst keratoconus based on maximum keratometry was selected as the Study Eye.

Any adverse events (AEs), suspected adverse events, and serious adverse events were recorded on the Adverse Event Report Form and in the patient's source documents. Laboratory, vital sign, or ECG abnormalities were recorded as AEs if medically relevant. The sponsor-investigator submitted a safety report to the review board no later than 15 calendar days after any suspected adverse reaction. Any unexpected fatal or life-threatening suspected adverse reactions was reported to the review board no later than 7 days after the sponsor-investigator's is made aware. Accidental or intentional overdose of the study drug or concomitant medication or discovery of pregnancy was reported to the Medical Monitor within 24 hours. Any AEs that led to a patient's withdrawal from the study were reported to the Medical Monitor within 30 days. In the case of an emergency, the Investigator could complete the subject treatment code breaking procedure. This was only done if awareness of the treatment had a direct impact on the subject's immediate medical management. The Medical Monitor was contacted prior to emergency unmasking or within 24 hours. The circumstances leading to unmasking of a subject were promptly communicated to the Sponsor and review board. A patient had the right to withdraw from the study at any time, for any reason, and without repercussion. The investigator had the right to withdraw a patient from the study in the event of an intercurrent illness, onset of pregnancy, adverse event (AE), treatment failure, or protocol violation. If a subject withdrew due to an AE(s), the reason for withdrawal was recorded as an adverse event. Subjects who failed to come to follow up visits and could not be contacted after 3 telephone calls followed by a certified letter were classified as "lost to follow-up".

Collected Data:

Corneal topography was obtained at every visit using the Oculus Pentecam. This device provided data for Maximum Central Keratometry (Kmax), Mean Central Keratometry (Kmean), Corneal Astigmatism, and Posterior Maximum Corneal Elevation.

The maximum central keratometry is a measure of the maximal corneal steepness and is a very commonly used in the diagnosis of keratoconus as well as monitoring and evaluating treatment effects. Normal Kmax is <49.00 diopters.

The mean central keratometry is a measure of the mean corneal steepness and anterior curvature. It is one of the measures of corneal topography which is the evaluation of the anterior curvature of the cornea. Normal Kmean is <47.20 diopters.

Corneal astigmatism is a measure of corneal irregularity leading to multiple focal points of light within the eye and impaired vision. Corneal astigmatism ranges greatly in magnitude and may be found in healthy patients to varying degrees, but it is also known to be present in keratoconus and worsens with disease progression. Keratoconus is the progressive and inferior bulging of the cornea. Therefore, corneal thickness is useful in diagnosis and disease or treatment monitoring. This was measured using the Oculus Pentecam at every visit. Central corneal thickness ranges from 472-651 micrometers and minimal thickness is normally >400 micrometers.

Intraocular pressure (IOP) above or below normal ranges may lead to pain or damage and may be affected by topical medications. IOP ranges from 8-21 millimeters of mercury.

An early sign of keratoconus is posterior thinning or "elevation". This measure is also useful in monitoring progression or treatment of the disease. Normal values are <17 micrometers.

The Ocular Response Analyzer (ORA) or Oculus Corvis were used at each visit. These are noncontact tonometers that use a puff of air to investigate the dynamic reaction and surface deformation of the cornea. These instruments provide an in vivo assessment of corneal biomechanics (i.e., resistance to corneal deformation) which may be used to monitor the progression and treatment of corneal diseases such as keratoconus. Normal values for measured parameters vary in the literature with no consensus currently. Analyzed variables from these machines include the corneal resistance factor (CRF) and corneal hysteresis from the ORA and stiffness parameter highest concavity (SP-HC), stress-strain index (SSI), and peak distance from the Oculus Corvis.

Mean Best Corrected Distance Visual Acuity (BCVA) is the vision patients achieve with proper correction of refractive error, i.e., wearing glasses. Uncorrected distance visual acuity (UCVA) is without correction. A standard Snellen Visual acuity chart was used to measure visual acuity at every visit.

Endothelial cells are located on the posterior surface of the cornea and are responsible for dehydration of corneal stroma ensuring its clarity. Damage to these cells and decrease in cell density may be caused by cytotoxic of topical medications. Endothelial cell count (EEC) was assessed at the Screening, Day 0, Week 6, and Week 26 (exit) visits with a specular microscope. EEC ranges from >1,500 to 3,500 cells per square millimeter.

Patients with discomfort and redness upon instillation was evaluated at each study visit. the Investigator recorded patient responses concerning perceived discomfort and redness following instillation away from the clinic. The case report form stated, "Did the patient experience discomfort immediately after using the assigned study drops?". Possible answers were "No" or "Yes". A "Yes" response was graded on a 5 point scale ranging from 1(slight discomfort) to 5 (very uncomfortable). Similarly, redness was measured with a 0 to 5 scales: 0 (white conjunctiva) to 5 (completely red conjunctiva).

Routine ophthalmic examination variables (external slit-lamp examination and dilated fundus examination) were also obtained performed.

Data Quality Assurance:

The progress of the study was monitored by on-site visits and with the use of telephone calls, e mails, and written communication between personnel at the study sites and the sponsor's representatives. Site personnel weighed assigned treatment bottles at each visit to monitor compliance. The Investigator allowed the clinical monitors or designees to inspect all completed case report forms, subject records (e.g., source documents), signed informed consent forms, records of study medication receipt, storage, and dispensation, and regulatory files related to this study. Monitoring and study management followed Good Clinical Practices. Patient data required for the study were recorded on paper case report forms completed during each office visit. The site sent copies of all case report forms and other study records to the sponsor in the form of PDF files. PDF files, with images of case report forms and printouts from the measuring equipment, were reviewed by the sponsor, indexed and archived in a Dropbox folder with limited access. All data were entered into Microsoft Excel spreadsheets by a masked clinical research monitor. Key efficacy and safety data was reviewed by a second masked individual and differences reconciled prior to unmasking. Some questionable Pentecam images were reviewed and validated by the masked medical monitor and invalid data was not included in the database. All original documents and source documentation were stored at the study site. All study documentation and source documents were made available upon request for inspection by authorized representatives from the sponsor or regulatory authorities.

The Data Safety Monitoring Committee:

The Committee included Balamurali Ambati, M.D. and Arturo Chayet, M.D. Types of adverse events monitored for and reviewed included, but were not limited to, endophthalmitis, increased IOP, cystoid macular edema, and retinal detachment. Study progress and safety reports were created by the monitoring committee. Findings of the monitoring committee were submitted to the review board after each meeting. In addition, the monitoring committee reviewed the data if any participant experienced a serious, unexpected adverse event. The investigator will retain all essential study documents, including ICFs, source documents, CRFs, and drug accountability records for at least 5 years following the completion or discontinuation of the study, or longer if a longer period is required by relevant regulatory authorities. Records will be destroyed in a manner that ensures confidentiality.

Determination of Sample Size:

This was a first-in-human study designed to assess safety and preliminary efficacy. No formal hypothesis testing, formal power calculations or sample size calculations were used to determine sample size. A sample size of up to 36 patients was targeted based on establishing a reasonable number of patients to provide adequate safety and preliminary efficacy information to proceed to the next phase of clinical development.

Statistical and Analytical Plan:

The Statistical Analysis Plan (SAP) was developed prior to the database lock for the primary and secondary efficacy and safety variables. This plan identified the primary endpoints, analysis and populations, and also the handling of missing data. The SAP was signed and approved before the data were unmasked for analysis. This is a proof of concept study to determine viability of topical copper sulfate eyedrops at slowing progression of keratoconus. The number of subjects enrolled is appropriate for a proof of concept study and not necessarily powered to demonstrate statistically significant differences between the groups. Reported statistics were descriptive (e.g., means, variance) and comparing results baseline measures with t-tests. Missing data for keratometry measures, Kmax, were imputed using a last z-score carried forward analysis. For the keratometry measure of interest, Kmax, additional analysis with a longitudinal linear mixed effects model was performed. Difference in slopes or means at 26 weeks will be compared between the IVMED-16Wk and Placebo group. Baseline measurements will be considered the average of measurements collected at the screening and day 0 visits if both are available. Data points that appear to be outliers will be investigated and will not be excluded from the listings unless the clinical investigator concludes the value is not clinically possible. If a clinically impossible outlier was found, two analyses were performed, one with and without clinically impossible data with footnotes to indicate the analyses. Slit-lamp findings and non-ophthalmic adverse events though collected were not analyzed for the topline analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Mild to moderate keratoconus and/or corneal ectasia post-LASIK or Photo-Refractive Keratectomy
2. Age 18 to 40
3. Minimum corneal thickness of > 350 microns
4. Maximum corneal keratometry of 45 D to 67 D
5. Absence of systemic comorbidities that pose a significant surgical risk
6. Absence of ocular comorbidities
7. Willing and able to comply with clinic visits and study-related procedures.
8. Provide signed informed consent

Exclusion Criteria:

1. Significant central corneal scarring or hydrops
2. Previous corneal surgeries
3. Presence of pre-existing glaucoma, uveitis, uncontrolled diabetic retinopathy, or prior ocular trauma or prior intraocular surgery.
4. Myopic degeneration with potential acuity less than 20/40 in the Study Eye.
5. Down's Syndrome, retinitis pigmentosa, Ehlers-Danlos Syndrome, osteogenesis imperfecta (or other collagen disorder) or Anton's Syndrome.
6. Prior retinal detachment involving the macula
7. Received a sub-Tenon's injection of corticosteroid within the past 6 months, or any intravitreal injection within the past 6 months in the study eye prior to Visit 1
8. Current use, or anticipated initiation during the study, of a systemic corticosteroid or an immunosuppressant agent by any route (oral, injectables)
9. History or current condition of substance or alcohol abuse within the past year
10. Participation in a clinical trial with use of any investigational drug or treatment within 30 days prior to Visit 1
11. Employee of the study site or their immediate families.
12. Pregnancy or planning to become pregnant.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-08 (Actual)

PRIMARY OUTCOMES:
Mean Maximum Central Keratometry (Kmax) | 26 weeks
  Change in maximum central keratometry after the assigned treatment was compared with baseline measures. This will be evaluated with and without z-score imputation. It will also be evaluated with a linear mixed effects model.
Number of Treatment-Emergent Adverse Events | 26 Weeks
  Treatment-emergent adverse events (TEAEs) were defined as events requiring additional treatments or cessation of the study article for which the date of onset was on or after the date of first dose of double-masked study drug at Day 0.
Mean Best Corrected Distance Visual Acuity (BCVA) | 26 Weeks
  Change in BCVA after the assigned treatment was compared with baseline measures.

SECONDARY OUTCOMES:
Mean Corneal Astigmatism | 26 Weeks
  Corneal astigmatism after the assigned treatment was compared with baseline measures.
Mean Central Keratometry (Kmean) | 26 Weeks
  The mean central keratometry after the assigned treatment was compared with baseline measures.
Mean Posterior Maximum Corneal Elevation | 26 Weeks
  Mean Posterior Maximum Corneal Elevation after the assigned treatment was compared with baseline measures.
Mean Endothelial Cell Count (ECC) | 26 Weeks
  Mean EEC after the assigned treatment was compared with baseline measures.
Percentage of patients with discomfort and redness upon instillation | 26 Weeks
  Percentage of patients with discomfort and redness upon instillation over the study period was reported.
Mean Corneal hysteresis | 26 weeks
  Mean Corneal hysteresis after the assigned treatment was compared with baseline measures with the Ocular Response Analyzer.
Mean Corneal resistance factor (CRF) | 26 weeks
  Mean Corneal resistance factor after the assigned treatment was compared with baseline measures with the Ocular Response Analyzer.
Mean Central Corneal Thickness (CCT) | 26 weeks
  The mean CCT after the assigned treatment was compared with baseline measures.
Mean Minimal Corneal Thickness | 26 weeks
  The mean Minimal Corneal Thickness after the assigned treatment was compared with baseline measures.
Mean Intraocular Pressure (IOP) | 26 weeks
  The mean IOP after the assigned treatment was compared with baseline measures.
Mean Uncorrected Visual Acuity (UCVA) | 26 Weeks
  The mean UCVA after the assigned treatment was compared with baseline measures.
Mean Stiffness parameter highest concavity (SP-HC) | 26 Weeks
  Mean SP-HC after the assigned treatment was compared with baseline measures with the Oculus Corvis.
Mean Stress-strain index (SSI) | 26 Weeks
  Mean SSI after the assigned treatment was compared with baseline measures with the Oculus Corvis.
Mean Peak distance | 26 Weeks
  Mean Peak distance after the assigned treatment was compared with baseline measures with the Oculus Corvis.

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Chayet, MD, Principal Investigator — Codet Vision Institute; Balamurali K. Ambati, MD, PhD, Study Director — iVeena Delivery Systems
Locations (1):
- Codet Vision Institute, Tijuana, Estado de Baja California, Mexico

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared in a journal publication.
Time Frame: Data will become available pending journal publication time frames.
Access Criteria: Data will be displayed in figures and tables and as supplemental files in the published journal and accessibility will depend on journal open access policies.

REFERENCES:
- [Background] Olivares Jimenez JL, Guerrero Jurado JC, Bermudez Rodriguez FJ, Serrano Laborda D. Keratoconus: age of onset and natural history. Optom Vis Sci. 1997 Mar;74(3):147-51. doi: 10.1097/00006324-199703000-00025. PMID 9159804
- [Background] Wagner H, Barr JT, Zadnik K. Collaborative Longitudinal Evaluation of Keratoconus (CLEK) Study: methods and findings to date. Cont Lens Anterior Eye. 2007 Sep;30(4):223-32. doi: 10.1016/j.clae.2007.03.001. Epub 2007 May 3. PMID 17481941
- [Background] Kymes SM, Walline JJ, Zadnik K, Sterling J, Gordon MO; Collaborative Longitudinal Evaluation of Keratoconus Study Group. Changes in the quality-of-life of people with keratoconus. Am J Ophthalmol. 2008 Apr;145(4):611-617. doi: 10.1016/j.ajo.2007.11.017. Epub 2008 Jan 28. PMID 18226798